CLINICAL TRIAL: NCT06596369
Title: Transcutaneous Spinal Cord Stimulation to Facilitate Recovery of Upper Extremity Function in Individuals With Stroke or Spinal Cord Injury - A Pilot Study
Brief Title: Transcutaneous Spinal Cord Stimulation for Upper Extremity Function
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Glenrose Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro001405596
Record Dates: First submitted 2024-06-06; First posted 2024-09-19 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries; Stroke
MeSH Terms: conditions — Spinal Cord Injuries; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tSCS + Rehab (Experimental): In this single arm study, individuals will receive transcutaneous spinal cord stimulation over the cervical spinal cord with upper extremity training utilizing the ReJoyce system.
  Interventions: Device: Transcutaneous spinal cord stimulation; Other: Upper extremity rehabilitation

INTERVENTIONS:
Device: Transcutaneous spinal cord stimulation — Continuous, sub motor threshold stimulation is delivered through surface electrodes placed over the cervical spine region.
Other: Upper extremity rehabilitation — Using the ReJoyce system individuals will engage in upper extremity rehabilitation.

SUMMARY:
Transcutaneous electrical stimulation (tcES) of the spinal cord has shown great promise in restoring upper extremity function after spinal cord injury (SCI). More recently, the use of invasive, epidural electrical stimulation of the spinal cord has also demonstrated promise in restoring upper extremity function post-stroke. However, the effect of stimulation parameters such as electrode configuration and stimulation frequency on excitability of the nervous system remains unknown preventing the opportunity to fully exploit this noninvasive stimulation paradigm. Additionally, the utility of noninvasive tcES in the stroke population remains unexplored. This project utilizes a comprehensive set of neurophysiological techniques, in combination with carefully chosen motor tasks, to directly link and assess the effects of stimulation parameters on neural excitability and upper extremity function during and following the delivery of cervical tcES in individuals with SCI and stroke. The fundamental knowledge gained from this project will ultimately improve the implementation of this novel and non-invasive neuromodulatory tool through an improved understanding of how tcES can facilitate recovery of function.

DETAILED DESCRIPTION:
In the first two aims of this study we explore the effects of stimulation configurations on neural excitability. Specifically we will explore the effects of electrode placement and stimulation frequency on measures of corticospinal and intracortical excitability. In the last aim of this study, individuals will participate in an interventional trial combining activity-based therapy with tcES. We will explore whether this intervention facilitated improvements in upper extremity function through clinical and neurophysiological assessments.

ELIGIBILITY:
Inclusion Criteria:

SCI cohort:

* individuals aged 18 to 75 years of age who have suffered a spinal cord injury
* cervical level injury (C3 to C8)
* at least 1-year post-injury
* for individuals taking medications for spasmolysis or muscle relaxation (e.g. oral baclofen, tizanidine, dantrolene, vigabatrin, gabapentin, or benzodiazepine), dose and regimen must be stable for at least 4 weeks prior to screening

Stroke cohort:

* individuals aged 18-75 years of age who have suffered any type of stroke resulting in upper extremity motor dysfunction with partially preserved motor function
* ≥ 6 months post-stroke
* At least 4 months since last BoNT injection for treatment of spasticity or any other condition or ≤ 2 months after study completion
* for individuals taking medications for spasmolysis or muscle relaxation (e.g. oral baclofen, tizanidine, dantrolene, vigabatrin, gabapentin, or benzodiazepine), dose and regimen must be stable for at least 4 weeks prior to screening

Exclusion Criteria:

* pregnant women
* aphasia or dysphasia
* spasticity grade Modified Ashworth Scale ≥ 3

Transcranial magnetic stimulation-specific exclusion criteria (both cohorts)

* participants with active or inactive implants including cardiac pacemakers, implantable defibrillators, ocular implants, deep brain stimulators, vagus nerve stimulator, and implanted medication pumps
* participants with conductive, ferromagnetic or other magnetic-sensitive metals implanted in their head
* participants with a history of seizures or epilepsy
* participants taking any medication which may reduce seizure threshold

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2029-09-14 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Spinal Excitability | Baseline, End of Intervention (2mths), 6-month follow-up (8mths)
  Changes in spinal excitability measured by stimulating the cervical spinal cord while recording muscle signals from upper extremity muscles will be assessed at the beginning and end of the interventional arm, and then 6 months following completion of the intervention.
Corticospinal excitability | Baseline, End of Intervention (2mths) and at 6-month follow-up timepoint (8mths)
  Changes in corticospinal excitability (using transcranial magnetic stimulation) will be assessed at the beginning and end of the interventional arm, and then 6 months following completion of the intervention.
Clinical assessment of UE function | Baseline, End of Intervention (2mths), and 6-month Follow-up (8mths).
  For SCI participants, the GRASSP assessment will be utilized to assess changes in upper extremity strength, sensation and function. In the stroke population, the ARAT, Fugl-Meyer tests will be utilized. In both patient groups, the arm and hand function test performed by the ReJoyce system will also be utilized.
Changes in Intracortical Excitability | Baseline, End of Intervention (2mths) and at 6-month follow-up timepoint (8mths)
  Changes in intracortical excitability utilizing paired-pulse transcranial magnetic stimulation protocols will be explored at baseline, end of the intervention period, and 6months following completion of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica D'Amico, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Glenrose Rehabilitation Hospital, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No
We do not plan to shared IPD with other researchers. Deidentified data may be shared with a data repository.